CLINICAL TRIAL: NCT06686784
Title: Using a Mentoring Afterschool Program to Improve Adolescent Mental Health and Physical Activity: A Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020498
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The crossover occurs after the first semester (end of Month 4). The study will occur with two middle schools.
  Months 1-4 Participants at "School A" (Arm 1) receive the Afterschool as Usual condition in the first semester. Participants at "School B" (Arm 2) receive the Afterschool Plus condition in the first semester.
  Months 5-8 Participants at "School A" (Arm 1) receive the Afterschool Plus condition in the second semester. and the participants at "School B" (Arm 2) receive afterschool as Usual condition in the second semester.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School A (Experimental): Middle school students at School A who participate in the after school program. They will receive after school as usual in months 1-4, followed by after school plus in months 5-8.
  Interventions: Behavioral: After School Plus
- School B (Experimental): Middle school students at School B who participate in the after school program. They will receive after school plus in months 1-4, followed by after school as usual in months 5-8.
  Interventions: Behavioral: After School Plus

INTERVENTIONS:
Behavioral: After School Plus — The afterschool program as usual runs M-H and consists of a variety of clubs from which middle school students chose to enroll for a semester (~4 months). Clubs are offered on either a M/W or T/H schedule. Students receive a snack in the cafeteria each day before attending their class.
  Afterschool plus is the same as "Afterschool as Usual" with the addition of young adult mentors. Following snack, mentors will lead students in a short emotion regulation exercise including physical activity and breathing exercises. Mentors will prompt students to identify how they are feeling and make connections between the activities they are doing and their mood and then do activities with students in each class. On T/H, ~4 mentors will lead a new "DiscoverU " club which is based on behavioral activation principles and spends more time helping students identify and do more activities that improve their mood. The class promotes physical activity as an important strategy for mental health.

SUMMARY:
Coming out of the COVID-19 pandemic many youth are experiencing declines in physical activity and worsening mental health (e.g., depression symptoms). These declines are exacerbated among underserved youth who experience greater barriers to health services and exposure to life stressors that put them at increased risk for impaired mental, emotional, and behavioral health. School-based afterschool programming is an important strategy to reach this population of youth and provides intervention at a time when youth are likely to otherwise be in environments not supportive of health. Further participation in extracurricular activities has been shown to be a protective factor for youth mental health. However, consistent with the Behavioral Theory of Depression, youth who are currently inactive and who have depression symptoms are unlikely to participate in afterschool programming on their own and likely require heightened positive reinforcement when they do attend to encourage retention. Given the high prevalence of youth who experience symptoms of depression and resource and staffing challenges faced by many schools, the level of support needed to engage students to consistently participate and benefit from afterschool programming is often beyond the capacity of school-based afterschool programs. In partnership with a local afterschool program for middle school students in a low resource community, the investigators developed an augmented version of the current afterschool program in which college students are trained to mentor and assist in the afterschool program, expanding the capacity of the afterschool program to engage students.

The mentoring intervention uses behavioral activation principles to help youth connect their behaviors with their mood and support youth to engage in behaviors that improve their mood, including physical activity. The main purpose of this study is to pilot the feasibility of the newly developed intervention.

DETAILED DESCRIPTION:
The proposed study builds from formative work in which the investigators developed an augmented version of an existing afterschool program in which college students are trained to mentor and assist in the afterschool program. Specifically, the mentoring intervention uses behavioral activation principles to help youth connect their behaviors with their mood and support youth to engage in behaviors that improve their mood, including physical activity. The main purpose of this study is to pilot the feasibility of the newly developed intervention. The study will use a modified, quasi-experimental crossover pilot trial design (n= 1 schools; 1 Afterschool program as usual and 1 After School Plus) conducted in partnership with St. Paul Public School District's school-based afterschool programming, "Flipside". School A will receive After School Plus in semester 1 and After School as Usual in semester 2. School B will receive After School as Usual in semester 1 and After School Plus in Semester 2. After School as Usual. The afterschool program as usual runs M-H and consists of a variety of clubs from which middle school students chose to enroll for a semester (~4 months). Clubs are offered on either a M/W or T/H schedule. Students receive a snack in the cafeteria each day before attending their class. During the After School as Usual condition, participants will not receive any extra intervention, but will participate in data collection using the same procedures and methodologies as the intervention schools.

After School Plus. After School Plus is the same as Afterschool as Usual with the addition of young adult mentors. Following snack, mentors will lead students in a short emotion regulation exercise including physical activity and breathing exercises. Mentors will prompt students to identify how they are feeling and make connections between the activities they are doing and their mood and then do activities with students in each class. On T/H, ~4 mentors will lead a new DiscoverU club which is based on behavioral activation principles and spends more time helping students identify and do more activities that improve their mood. The class promotes physical activity as an important strategy for mental health. Recruitment. Adolescents will be invited to participate in the study when they enroll in the afterschool program. The investigators will work closely with the site lead and teacher at each school assigned to help us with recruitment and retention. Adolescents can participate in the afterschool program without participating in the study (i.e., data collection).

Parents will need to provide written parental consent and students provide written assent before a student can enroll in the study. Because students can enroll in afterschool program at any time over the year, we will allow study enrollment on an ongoing basis through February 2025. Mentors will be recruited by emailing a description of the mentor opportunity to various student organizations and professors to share with their classes. This study targets courses with large class sizes. The study will also post flyers describing the opportunity across campus.

Promising candidates based on their application will be invited to group information sessions at which the research team observes their interactions in a group setting and provides information about the role. Interested candidates are asked to schedule a one- on-one interview. Mentors can receive class credit for mentoring. We previously used these strategies in the proof-of-concept study to recruit a diverse group of mentors, reflective of many majors and colleges. Data Collection. Primary data collection will include process data (e.g., attendance) and pre, midpoint, and post surveys (October, December, and April) among adolescents and mentors. Surveys will assess constructs including depressive symptoms, anxiety symptoms, behavioral activation, and emotion regulation. Additionally, approximately 75-80% of adolescent participants will provide accelerometry data to measure the amount and intensity of physical activity they do during the afterschool program

ELIGIBILITY:
Student Inclusion Criteria:

* Any 6th , 7th , or 8th grade student who is enrolled in their after school plus program at a participating middle school

Parent/Guardian Inclusion Criteria:

* Any parent of a student who is enrolled in the study is eligible to participate.

Mentor Inclusion Criteria:

* Any mentor in the after school plus program is eligible to participate.

Staff Member Inclusion Criteria:

* Any staff member affiliated with the after school program at a participating middle school

Exclusion Criteria:

* Have a substantial cognitive impairment that would prevent the completion of data collection activities.

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
intervention feasibility | 4 months
  This will be measured by participant semester 1 rate of attendance at the after school program (i.e., the number of days attended divided by the number of days the class(es) the student was signed up for were offered in semester 1)
intervention feasibility | 8 months
  This will be measured by participant semester 2 rate of attendance at the after school program (i.e., the number of days attended divided by the number of days the class(es) the student was signed up for were offered in semester 2)

SECONDARY OUTCOMES:
Depression symptoms | Baseline
  Will be measured using PHQ-8
Depression symptoms | 4 months
  Will be measured using PHQ-8
Depression symptoms | 8 months
  Will be measured using PHQ-8
Activity level in after school program | 4 months
  Accelerometry measured 2 days per semester at randomly selected intervals per class
Activity level in after school program | 8 months
  Accelerometry measured 2 days per semester at randomly selected intervals per class

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hendel, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States